CLINICAL TRIAL: NCT06338696
Title: Thailand Transthyretin Amyloid Cardiomyopathy Registry
Brief Title: Thailand ATTR-CM Registry
Status: Recruiting | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Rungroj Krittayaphong, Professor, Mahidol University
Other Study IDs: COA-CREC070/2023
Record Dates: First submitted 2024-03-14; First posted 2024-04-01 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Transthyretin Amyloid Cardiomyopathy (ATTR-CM)
Keywords: Transthyretin amyloid cardiomyopathy (ATTR-CM); Heart Failure; Cardiomyopathy
MeSH Terms: conditions — Heart Failure; Cardiomyopathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ATTR Cardiomyopathy: Patients diagnosed with ATTR-CM (Transthyretin cardiomyopathy)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The investigators of this registry aim to study the natural history, clinical presentation, characteristics, and imaging findings of patients diagnosed with ATTR amyloidosis in Thailand longitudinally. This will enable the investigators to study this disease in depth. With a better understanding, the investigators can aim to develop early screening programs for at-risk patients, raising awareness among non-cardiologists. As amyloid-specific therapies have now become available in Thailand, the findings of this registry can be helpful for epidemiological studies in Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* All patients diagnosed with ATTR-CM (Transthyretin cardiomyopathy) who have either symptomatic or asymptomatic must have evidence of cardiac involvement by echocardiogram as defined by left ventricle wall thickness of ≥ 12 mm and with at least one of the following criteria:
* Positive scintigraphy by 99mTC-DPD [99mTC-3,3-diphosphono-1,2-propano-dicarboxylic acid] or 99mTC-PYP [Pyrophosphate] or 99mTC-HMDP [hydroxymethylene diphosphate] with Perugini grade ≥ 2 and/or H/CL (heart to contralateral lung) ratio > 1.5
* Positive scintigraphy by 99mTC-DPD [99mTC-3,3-diphosphono-1,2-propano-dicarboxylic acid] or 99mTC-PYP [Pyrophosphate] or 99mTC-HMDP [hydroxymethylene diphosphate] with Perugini grade 1 and positive cardiac biopsy tissue confirmed which Congo red stain ≥ 4 sites
* Positive scintigraphy by 99mTC-DPD [99mTC-3,3-diphosphono-1,2-propano-dicarboxylic acid] or 99mTC-PYP [Pyrophosphate] or 99mTC-HMDP [hydroxymethylene diphosphate] with Perugini grade 1 with positive non-cardiac biopsy tissue confirmed by Congo red stain
* Abnormalities on CMR (Cardiac MRI) [Subendocardium LGE (late gadolinium enhancement) and/or elevated native T1 value and/or increased extracellular volume (ECV > 0.4)] with positive non-cardiac and/or cardiac tissue biopsy confirmed by Congo red stain

Exclusion Criteria:

* Diagnosed with amyloidosis caused by proteins other than transthyretin (light chain Amyloidosis, etc.)
* Diagnosed with secondary amyloidosis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with ATTR-CM,Transthyretin cardiomyopathy, who have either symptomatic or asymptomatic.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of death | 3 years
Rate of heart failure hospitalization | 3 years

SECONDARY OUTCOMES:
Transthyretin (ATTR) amyloidosis medication | 3 years
  Rate of use and rate of adverse effect of Transthyretin (ATTR) amyloidosis medication

CONTACTS AND LOCATIONS:
Overall Officials: Rungroj Krittayaphong, MD, FESC, FACC, Principal Investigator — Division of Cardiology, Department of Medicine, Siriraj Hospital, Mahidol University
Locations (8):
- Thailand (8):
  - Faculty of Medicine at Chulalongkorn University, Bangkok
  - Faculty of Medicine Ramathibodi hospital, Mahidol University, Bangkok
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Faculty of Medicine Chiang Mai University, Chiang Mai
  - Queen Sirikit Heart Center of The Northeast, Khon Kaen
  - Faculty of Medicine, Thammasat University, Pathum Thani
  - Prince of Songkla University, Songkhla